CLINICAL TRIAL: NCT04152746
Title: Periostin Levels in Children With Adenoid Hypertrophy
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: 8/8.11.04.2018
Record Dates: First submitted 2019-10-23; First posted 2019-11-05 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Adenoid Hypertrophy
Keywords: Adenoid Hypertrophy; Periostin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Adenoid tissue and blood samples were collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adenoid group: Periostin levels in the adenoid group
  Interventions: Other: Periostin level
- Control Group: Periostin levels in the control group
  Interventions: Other: Periostin level

INTERVENTIONS:
Other: Periostin level — The serum periostin levels were planned to compare between the serum samples that were obtained from the two groups. The evaluation of the periostin levels of adenoid tissue and normal healthy mucosa were also planned.

SUMMARY:
Periostin is a matricellular protein that has been shown to be a marker of Type 2 inflammation associated with airway eosinophilia. Matricellular proteins are highly expressed at sites of injury or inflammation. Periostin involves tissue fibrosis and remodeling in the nasal mucosa in some of the otolaryngologic diseases. The up-regulation of periostin expression has been shown in allergic rhinitis, chronic rhinosinusitis with nasal polyps , and aspirin intolerant asthma. In the light of these findings the investigators aimed to evaluate the relation between adenoid hypertrophy and periostin levels.

DETAILED DESCRIPTION:
A total of 40 patients-age ranged between 2 and 12 years- were planned to enroll in the study prospectively. Patients that were scheduled to undergo adenoidectomy were included in the study group (adenoid group). The control group comprised of 20 healthy children who had previously been treated for anemia in the out-patient clinic of the Pediatrics Department and were clinically healthy with normal complete blood cell counts at their follow-up visits.

Serum samples were obtained from the two groups. The samples were centrifuged at 1500 g for 5 minute and stored in -80 oC for later analysis of periostin levels. Adenoid tissue and normal mucosal tissue samples were obtained from the adenoidectomy patients and stored in -80 oC for later homogenization and measurement of periostin levels.

ELIGIBILITY:
Inclusion Criteria:

* The patients that were scheduled for adenoidectomy
* Healthy subjects that had not any kind of allergy, adenoid hypertrophy symptoms

Exclusion Criteria(for adenoid group):

* The subjects that had any kind of corticosteroid treatment 1 month prior to surgery, and antihistaminic treatment 2 weeks prior to surgery

Exclusion Criteria(for control group):

* To have allergic rhinitis symptoms
* To have high total IgE levels
* To have positive skin prick test
* To have acute respiratory tract infection
* To have asthma To have any kind of endocrin disease

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients that were scheduled to undergo adenoidectomy were included in the study group (adenoid group). The control group comprised of healthy children who had previously been treated for anemia in the out-patient clinic of the Pediatrics Department and were clinically healthy with normal complete blood cell counts at their follow-up visits.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-02-02 (Actual)

PRIMARY OUTCOMES:
Serum Periostin level | 1 month
  Serum periostin levels of the adenoid group and control group will be compared.
Adenoid tissue Periostin level | 1 month
  Periostin levels of the adenoid tissue and normal mucosal healthy tissue will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Nazan Degirmenci, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No